CLINICAL TRIAL: NCT00467766
Title: Combining a Caregiver Intervention With Aricept Treatment for Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Organization: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IA0114
Record Dates: First submitted 2007-04-27; First posted 2007-05-01 (Estimated); Last update posted 2007-05-07 (Estimated); Status verified 2007-05

CONDITIONS: Alzheimer Disease; Caregivers
Keywords: dementia; Counseling
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Counseling; Palliative Care; Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Psychosocial information, counseling, and support
Drug: Donepezil (Aricept)

SUMMARY:
A unique multinational study was conducted simultaneously in the USA, England and Australia. The goals of the study were to answer two questions: Does psychosocial support for the family enhance the effectiveness of drug treatment for Alzheimer's disease? Is the added value of psychosocial support the same in all 3 countries?

DETAILED DESCRIPTION:
This study is a single-blind prospective randomized trial with 150 patient/caregiver pairs (50 in each country). Eligibility criteria at baseline require that the primary caregiver is the spouse of the patient; the patient must have a diagnosis of AD, be in the in mild to moderate stage of dementia, be living with the caregiver, and be willing to take Donepezil (Aricept). These participants were randomly assigned to one of two groups: in one group, the intervention consists of drug treatment for the patient plus psychosocial intervention for the caregiver; in the other group the intervention consists solely of drug treatment for the patient.

The intervention for the caregiver consists of 5 scheduled individual and family counseling sessions within 3 months of baseline, and unlimited consultations on request. Assessments were conducted every 3 months for the first year and every 6 months for a second year. There are 3 sources of data: an interview of the caregiver by an independent rater, an assessment of the patient, and a count of the amount of medication used. Thus we will be able to assess the effect of adding counseling to medication for the caregiver, for the patient, and on compliance with medication use.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with mild to moderate stage Alzheimer's disease and their spouse caregivers

Exclusion Criteria:

* Severe psychological or physical illness
* Unwillingness by either spouse to participate in all aspects of the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 1999-07; Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Caregiver: Changes in depression, measured with the Beck Depression Inventory | every 3 months for the first year, and every 6 months for the second year
Caregiver: Changes in social support satisfaction, measured with the Stokes Social Network Scale | every 3 months for the first year, and every 6 months for the second year
Patient: Changes in cognition measured by ADAS-cog | every 3 months for the first year, and every 6 months for the second year
Patient: Changes in abilities with activities of daily living measured by ADCS-ADL | every 3 months for the first year, and every 6 months for the second year

SECONDARY OUTCOMES:
Caregiver: Changes in reactions to patient behavior, physical health, family conflict and sense of mastery | every 3 months for the first year, and every 6 months for the second year
Patient: Time to nursing home placement

CONTACTS AND LOCATIONS:
Overall Officials: Mary S. Mittelman, DrPH, Principal Investigator — NYU School of Medicine
Locations (3):
- Aging and Dementia Research Center, Silberstein Institute, NYU School of Medicine, New York, New York, United States
- Prince of Wales Hospital, Randwick, New South Wales, Australia
- University of Manchester, Division of Psychiatry, Manchester, United Kingdom

REFERENCES:
- [Background] Mittelman MS, Haley WE, Clay OJ, Roth DL. Improving caregiver well-being delays nursing home placement of patients with Alzheimer disease. Neurology. 2006 Nov 14;67(9):1592-9. doi: 10.1212/01.wnl.0000242727.81172.91. PMID 17101889
- [Background] Mittelman MS, Roth DL, Coon DW, Haley WE. Sustained benefit of supportive intervention for depressive symptoms in caregivers of patients with Alzheimer's disease. Am J Psychiatry. 2004 May;161(5):850-6. doi: 10.1176/appi.ajp.161.5.850. PMID 15121650
- [Background] Jang Y, Clay OJ, Roth DL, Haley WE, Mittelman MS. Neuroticism and longitudinal change in caregiver depression: impact of a spouse-caregiver intervention program. Gerontologist. 2004 Jun;44(3):311-7. doi: 10.1093/geront/44.3.311. PMID 15197285
- [Background] Roth DL, Mittelman MS, Clay OJ, Madan A, Haley WE. Changes in social support as mediators of the impact of a psychosocial intervention for spouse caregivers of persons with Alzheimer's disease. Psychol Aging. 2005 Dec;20(4):634-44. doi: 10.1037/0882-7974.20.4.634. PMID 16420138